CLINICAL TRIAL: NCT03720561
Title: EValuate Ibrutinib Retention iN Chronic Lymphocytic Leukemia Patients Treated in a rEal World Setting - EVIdeNCE
Brief Title: A Study to Evaluate Ibrutinib Retention in Chronic Lymphocytic Leukemia Participants Treated in a Real World Setting
Acronym: EVIdeNCE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108517; 54179060CLL4013 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Group: Ibrutinib Treatment: Participants will not receive any intervention as a part of this study. This study will collect retrospective and prospective real-world data to describe retention rates for participants of chronic lymphocytic leukemia (CLL) receiving ibrutinib in routine Italian clinical practice over a 2-year follow-up period. Participants with CLL who have started ibrutinib treatment within 3 months before enrollment visit or in case ibrutinib was prescribed before or on the enrollment day as per routine clinical practice within the 30 days after enrollment visit will be included in the study. The primary data source for this observational study will be the medical records of each enrolled participant, as well as questionnaires concerning quality of life and treatment adherence. Data will be collected every 3 months for the first year and every 6 months for the second year during prospective period.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants in this observational study with confirmed diagnosis of CLL receiving ibrutinib in routine clinical practice settings will be observed approximately for 3 years.

SUMMARY:
The purpose of this study is to describe the 2-year retention rate of ibrutinib treatment for chronic lymphocytic leukemia (CLL) in Italian routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL) requiring treatment (iwCLL [International Workshop on Chronic Lymphocytic Leukemia] criteria)
* If alive, must sign an Informed Consent Form (ICF) allowing data collection and source data verification in accordance with Italian requirements
* Participants with one of the following characteristics: a) Participants starting ibrutinib treatment according to the summary of product characteristics (SmPC) at enrolment or within 30 days starting from informed consent signature, as per routine clinical practice and independently of this non-interventional study; OR b) Participants who have started ibrutinib within 3 months before enrollment, according to the SmPC, as per routine clinical practice and independently of this non- interventional study (including also participants who, by the time of enrollment, are not receiving ibrutinib)
* If alive, must be able to read and write in Italian and to understand and sign the ICF

Exclusion Criteria:

* Currently enrolled in any interventional clinical trial
* Currently enrolled in observational studies sponsored or managed by Janssen company
* Treated with any investigational compound or any invasive investigational medical device within 30 days before start of ibrutinib treatment
* Having contraindications to ibrutinib use as described in the SmPC
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes participants who already started ibrutinib treatment within 3 months before enrollment visit or was prescribed ibrutinib before or on the enrollment day as per routine clinical practice - within the 30 days after enrollment visit. Along with alive participants, also deceased or untraceable participants who are eligible based on the selection criteria, their data will be collected for the evaluation of primary objective of the study.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Retention Rate of Ibrutinib | Approximately up to 2 years
  The retention rate is defined as the ratio of the number of participants taking ibrutinib over the number of participants at risk. The retention rate of ibrutinib treatment for (Chronic lymphocytic leukemia) CLL in Italian routine clinical practice will be measured.

SECONDARY OUTCOMES:
Number of Participants Requiring Dose Modifications | Approximately up to 2 years
  Number of CLL participants with at least one ibrutinib treatment dose modification (that is, increase/decrease) will be reported.
Overall Response Rate (ORR) | Approximately up to 2 years
  The ORR will be calculated as the proportion of participants who achieve either complete response (CR), partial response (PR) or partial response with lymphocytosis, as assessed by the participating physician. The ORR in CLL participants as per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria is defined as normal circulating lymphocyte count during CR and decrease by greater than or equal to (>=) 50 percent (%) during PR.
Time to Best Response | Approximately up to 2 years
  Time to best response is defined as the time from start of ibrutinib therapy until best objective response. Best response will be evaluated based on the following generally accepted algorithm: complete response greater than (>) partial response > partial response with lymphocytosis > stable disease > progressive disease.
Time to Treatment Discontinuation(TTD) | Approximately up to 2 years
  Time to treatment discontinuation (TTD) will be calculated as the difference between ibrutinib initiation date and ibrutinib permanent discontinuation date.
Time to Next Therapy (TTNT) | Approximately up to 2 years
  The TTNT will be calculated as the difference between ibrutinib initiation date and initiation date of the first next therapy for CLL.
Progression Free Survival (PFS) | From the date of assignment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 2 years
  PFS is defined as the duration from date of ibrutinib initiation to date of disease progression (PD [according to the physician's evaluation]) or death from any cause. PD is defined as >= 50% increase in circulating lymphocyte count as per iwCLL criteria.
Overall Survival (OS) | From the date of assignment until the date of death from any cause, whichever comes first, assessed up to 2 years
  The OS in CLL participants will be measured and reported from start of ibrutinib therapy to the date of death (all-cause mortality); and from diagnosis to the date of death.
Number of Participants with Clinically Significant Change in Hematologic Parameters | Approximately up to 2 years
  Number of participants with change in hematologic parameters (complete blood count, hemoglobin, leukocyte count, lymphocyte count, neutrophil count, platelet count) will be determined.
Number of Participants with Clinically Significant Change in Biochemistry Parameters | Approximately up to 2 years
  Number of participants with clinically significant change in biochemistry parameters (including lactate dehydrogenase [LDH] and creatinine clearance) will be determined.
Change from Baseline in Immunoglobulin levels | Baseline up to 2 years
  Changes in the immunoglobulin levels from baseline will be reported.
Number of Participants with at least one Clinical Significant Characteristics | Approximately 2 years
  Number of participants with at least one of the following conditions: lymphadenopathy, hepatosplenomegaly, bone marrow involvement, or B-symptoms as provided will be reported.
Number of Participants with Each Grade of Eastern Cooperative Oncology Group (ECOG) Performance Status Score | Approximately up to 2 years
  ECOG performance status is a standard criterion for measuring how the disease impacts daily living abilities. It describes the level of functioning in terms of the ability to care for oneself, daily activity, and physical ability (walking, working, etc). ECOG performance status score ranges from Grade 0 to 5: 0) Fully active and performances without restriction, 1) Restricted in physically strenuous activity, 2) Ambulatory and capable of all self-care but unable to carry out any work activities, 3) Capable of only limited self-care and confined to bed or chair more than 50% of waking hours, 4) Completely disabled, and 5) Dead.
Percentage of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and Special Situations | Approximately up to 2 years
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Percentage of participants with AEs, all serious AEs, and all special situations (for example, medication error, overdosing, abuse, lack of effect, unexpected benefits following exposure to ibrutinib) will be reported.
Health-Related Quality of Life as Measured by European Quality of Life-5 Dimensions; 5 Levels Questionnaire (EQ-5D-5L) | Approximately up to 2 years
  The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Health-Related Quality of Life as Measured by European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) Scores | Approximately up to 2 years
  EORTC QLQ-30 designed to measure cancer patients' physical, psychological and social functions. It is composed of multi-item scales (physical, role, social, emotional and cognitive functioning) and single items (pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life); high scores on the global and functional scales but low scores on the symptom scales indicate good QOL. QLQ-C30 has four-point scales for the first five items. These are coded with the same response categories as items 6 to 28, namely "Not at all", "A little", "Quite a bit" and "Very much." For items 29 and 30, a seven-point scale (ranging from 1 = "Very Poor" to 7 = "Excellent") rates overall health and overall quality of life.
Medical Resource Utilization | Approximately up to 2 years
  Number of medical care encounters and treatments (including physician or emergency room visits, tests and procedures, and medications, surgeries and other procedures [such as computerized tomography {CT}, x-ray]) will be reported.
Duration of Hospitalization | Approximately up to 2 years
  Duration of hospitalization is defined as number of days from the day of admission to discharge (total days length of stay), including duration by wards (for example, intensive care unit).
Duration of Medical Care Encounters | Approximately up to 2 years
  Duration of medical care encounters, including surgeries, and other selected procedures (inpatient and outpatient) will be reported.
Number of Participants Requiring Blood and Platelets Transfusions | Approximately up to 2 years
  Number of participants requiring blood and platelets transfusions will be reported.
Number of Participants Requiring Erythropoietin and Growth Factor Administrations | Approximately up to 2 years
  Number of participants requiring erythropoietin and growth factor administrations will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (39):
- Italy (39):
  - Ospedali Riuniti Di Ancona, Ancona
  - U.O.C. Ematologia e Terapia Cellulare Ospedale C e G Mazzoni, Ascoli Piceno
  - U.O. Ematologia con Trapianto- AOU Policlinico di Bari, Bari
  - U.O. Ematologia Istituto Tumori Giovanni Paolo II, Bari
  - S.C. Ematologia e CTMO P.O. Businco A.O. Brotzu, Cagliari
  - AORN Sant'anna e San Sebastiano, Caserta
  - Div.Clinicizzata EmatologiaconTrapiantodi MidolloOsseo P.O.Rodoligo AOUPoliclinico-Vittorio Emanuele, Catania
  - S.O.C. Ematologia P.O. Ciaccio A.O. Pugliese-Ciaccio, Catanzaro
  - Azienda Ospedaliero Universitaria di Ferrara, Cona
  - S.C. Ematologia Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Unità Funzionale di Ematologia Azienda ospedaliero-universitaria Careggi, Florence
  - S.C. Ematologia A.O.U. Ospedali Riuniti, Foggia
  - Ematologia Ospedale San Martino, Genova
  - U.O.C. Ematologia Ospedale V. Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - U.O.C. Ematologia Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Programma di ricerca strategica sulla LLC Ospedale San Raffaele, Milan
  - Divisione ematologia Grande Ospedale Metropolitano Niguarda, Milan
  - Division of Hematology, Cardarelli Hospital, Napoli
  - U.O.C. Ematologia e Trapianti di midollo A.O.U. Federico II, Napoli
  - Ospedale San Francesco, Nuoro
  - U.O.C. Ematologia e Immunologia Clinica Azienda Ospedaliera Padova, Padua
  - U.O. Ematologia ed Oncologia Ospedale A. Tortora, Pagani
  - Ospedale 'Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - S.C. Ematologia A.O.U. Santa Maria della Misericordia, Perugia
  - UOSD Centro diagnosi e terapia dei linfomi Ospedale Santo Spirito, Pescara
  - U.O.C. Ematologia Ospedale S. Maria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - DH Oncoematologia Policlinico Tor Vergata, Roma
  - Università di Roma 'La Sapienza' - Ospedale Umberto 1°, Roma
  - Ematologia Fondazione Univ. Policlinico Gemelli Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliera Sant Andrea, Roma
  - UO Oncologia ed Ematologia Istituto Clinico Humanitas, Rozzano
  - U.O.C. Ematologia e Trapianti Cellule Staminali Emopoietiche AOU S.Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Ospedale 'Casa Sollievo della Sofferenza' - U.O. Ematologia-, San Giovanni Rotondo
  - Azienda Ospedaliera 'Santa Maria', Terni
  - S.C. Ematologia U A.O.U. Citta della Salute e della Scienza P.O.Molinette, Torino
  - U.O. Ematologia Ospedale San Bortolo, Vicenza